CLINICAL TRIAL: NCT02663661
Title: Insulin-Glucose-Glucagon Network: Defining a Type 1 Diabetes Progression Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leon Farhi, PhD, Principal Investigator, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18568; DP3DK106907-01 (NIH)
Record Dates: First submitted 2015-12-07; First posted 2016-01-26 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1 (T1DM); TrialNet; Pathway to Prevention (PTP); First and second degree relatives of persons with T1DM; Insulin-glucagon-glucose (IGG); Immunological risk to develop T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autoantibody negative subjects (Other): Subjects who are relatives of persons with T1DM and have tested negative for autoantibodies will have a Metabolic Challenge Admission followed by a CGM home test.
  Interventions: Procedure: Metabolic Challenge Admission; Other: CGM home test
- One autoantibody subjects (Other): Subjects who are relatives of persons with T1DM and have tested positive for one autoantibody will have a Metabolic Challenge Admission followed by a CGM home test..
  Interventions: Procedure: Metabolic Challenge Admission; Other: CGM home test
- Two or more autoantibody subjects (Other): Subjects who are relatives of persons with T1DM and have tested positive for two or more autoantibodies will have a Metabolic Challenge Admission followed by a CGM home test..
  Interventions: Procedure: Metabolic Challenge Admission; Other: CGM home test

INTERVENTIONS:
Procedure: Metabolic Challenge Admission — A ten hour clinical test involving drinking a liquid mixed meal followed four hours later by the induction of hypoglycemia with intravenous insulin administration.
Other: CGM home test — A home study starting immediately after the clinical test during which participants will wear a continuous glucose monitor (CGM) for one week.

SUMMARY:
The type 1 Diabetes (T1D) TrialNet Pathway To Prevention (PTP) Study assesses and recruits at-risk subjects into clinical trials aimed at preventing the development of full blown T1D. Thousands of first and second degree relatives of persons with T1D are screened for autoimmune abnormalities and positive subjects are followed with metabolic and autoantibody tests. The investigators' ancillary study us designed to test whether characterization of the insulin- glucose-glucagon (IGG) interactions in participants in the PTP study can provide new information about the early stages of the disease. When completed, this study will improve the understanding of the pathogenesis of the early stages of T1D and provide new quantitative tools for prediction and evaluation of insulin-glucagon-glucose interactions relevant to individuals at risk for developing T1D, thereby enabling future preventive intervention trials.

DETAILED DESCRIPTION:
The goal of the proposed ancillary studies is to establish whether characterization of the insulin-glucagon-glucose (IGG) interactions in first and second degree relatives of patients with type 1 diabetes (T1D) can provide new information about the pathogenesis, prediction, and progression of the early stages of the disease. The project will enroll individuals from the "Living Biobank" of the TrialNet Pathway to Prevention (PTP) study who are phenotyped with respect to a variety of risk factors, including immunological abnormalities. To the best of available knowledge, the IGG relationships in general and the glucagon phenotype in particular have not been studied in this population. It is known, however, that in T1D the release of glucagon is altered, which is manifested by abnormal postprandial suppression and defective response to hypoglycemia. Several reports indicate that glucagon becomes dysregulated prior to the development of T1D, but comprehensive studies aiming to understand in detail the insulin-glucagon co-dynamics in people at risk for T1D have never been performed.

Thus, the goal now is to expand the investigators' existing methodology and transfer expertise in clinical testing and analysis of the IGG system to characterize the IGG interactions in individuals at risk for developing T1D.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 12 to 45 years old which have a brother, sister, child, or parent with type 1 diabetes, or
* Individuals 12-20 years old who have have a cousin, aunt, uncle, niece, nephew, half-brother, half-sister, or grandparent with type 1 diabetes.

Exclusion Criteria:

* Have diabetes already (type 1 or type 2)
* Have a medical condition or being been treated with medications that might interfere with the study

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that immunological abnormalities are associated with abnormally high glucagon responses to a meal and reduced glucagon responses to insulin induced hypoglycemia. | Approximately 10 hours
  To address this aim, subjects in all three groups which are at different level of immunological risk to develop T1D will undergo a single 10-hour clinical test consisting of a mixed meal drink followed by insulin-induced hypoglycemia (Metabolic Challenge) to estimate their postprandial and counterregulatory glucagon responses.

SECONDARY OUTCOMES:
Correlate metrics derived from a minimally-invasive Continuous Glucose Monitor (CGM) home test with glucagon responses to a meal and hypoglycemia measured in the hospital. | Seven days
  Subjects will undergo a CGM home test. They will wear a CGM for a week at home, keep a meal diary, and ingest a mixed meal of known amount with a subsequent collection of urine sample. A novel mathematical methodology will be used to extract from the field data estimates of the glucagon responses to a meal and to a decline in blood glucose levels. It will be then tested whether this estimates correlate to the glucagon responses measured in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Farhy, PhD, Principal Investigator — UVA Center for Diabetes Technology; Sue A Brown, MD, Principal Investigator — UVA Center for Diabetes Technology
Locations (1):
- University of Virginia, Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Montaser E, Breton MD, Brown SA, DeBoer MD, Kovatchev B, Farhy LS. Predicting Immunological Risk for Stage 1 and Stage 2 Diabetes Using a 1-Week CGM Home Test, Nocturnal Glucose Increments, and Standardized Liquid Mixed Meal Breakfasts, with Classification Enhanced by Machine Learning. Diabetes Technol Ther. 2023 Sep;25(9):631-642. doi: 10.1089/dia.2023.0064. Epub 2023 Jun 15. PMID 37184602